CLINICAL TRIAL: NCT06487039
Title: A Randomization, Double-blind, Parallel, Multicenter-Phase 2a Trial to Evaluate the Safety and Efficacy of EB-203 in Patients With Neovascular Age-related Macular Degeneration
Brief Title: Trial to Evaluate the Safety and Efficacy of EB-203 in Patients With Neovascular Age-related Macular Degeneration
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: EyebioKorea, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EB-203-201
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Neovascular Age-related Macular Degeneration (nAMD)
Keywords: nAMD; eye

STUDY DESIGN:
Intervention Model Description: Group A: EB-203 2% QID Group B: EB-203 4% QID
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): EB-203 2% QID
  Interventions: Drug: EB-203
- Group B (Experimental): EB-203 4% QID
  Interventions: Drug: EB-203

INTERVENTIONS:
Drug: EB-203 — Subjects will receive EB-203 according to the following dosage and administration method for each treatment group.

SUMMARY:
Trial to Evaluate the Safety and Efficacy of EB-203 in Patients with Neovascular Age-related Macular Degeneration.

The purpose of this study is to primarily investigate the safety and tolerability of EB-203 by dose in patients with neovascular Age-related Macular Degeneration (nAMD), and to secondarily evaluate the clinical efficacy. Subject to Adults aged 50 years or older and Neovascular age-related macular degeneration (nAMD)

DETAILED DESCRIPTION:
This study is a double-blind, parallel, multicenter-phase 2a study to evaluate the safety and efficacy of EB-203 in patients with nAMD.

Subjects who have been informed about the study and have voluntarily agreed to sign to participate in the study will be screened.

Final subjects who meet the inclusion/exclusion criteria will be randomized in a 1:1 ratio into Group A(EB-203 2%, 4 times a day) and Group B (EB-203 4%, 4 times a day).

Randomization will be performed using the study institution (hereinafter "institution") as a stratification factor.

Subjects will receive the investigational products according to the group to which they are randomized.

Safety and tolerability will be assessed for 12 weeks after randomization. Efficacy will be assessed at Weeks 4, 8, and 12. In addition, subjects will be monitored by visiting the institution 4 weeks after the last dose of the investigational product (Visit 8).

If a subject meets the criteria for the administration of rescue medication at Visit 3 (Week 2), he/she will be withdrawn from the study.

From Visit 4 (Week4), subjects may be withdrawn from the study based on the withdrawal criteria for each visit or the criteria for the administration of rescue medication.

If a subject who meets the criteria for the administration of rescue medication for each visit is withdrawn from the study, he/she will be administered the anti-VEGF drug aflibercept (product name: Eylea Injection®) once (intraocular injection).

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 50 years or older
2. Subjects with a best corrected visual acuity (BCVA) score between 25 and 73, measured by the Early Treatment of Diabetic Retinopathy Study(ETDRS) chart, at a distance of 4 m during the screening (equivalent to 20/40 to 20/320 in the Snellen chart)
3. Subjects who voluntarily signed the informed consent form (ICF) after receiving the information on this study

Exclusion Criteria:

1. Subjects with confirmed nAMD requiring standard treatment in both eyes (however, dry AMD in the non-study eye may be enrolled)
2. Subjects who have received ocular or systemic treatment, such as photodynamic therapy (PDT) or laser photocoagulation, or have undergone a surgical operation for nAMD (however, health functional foods, vitamin supplements, etc., are excluded)
3. Subjects whose study eye has been treated with anti-vascular endothelial growth factor (anti-VEGF) drugs (e.g. ranibizumab, bevacizumab, aflibercept, etc.) or a combination therapy for the treatment of nAMD prior to screening
4. Subjects who have received intravitreal treatment using steroids
5. Subjects who have a subretinal hemorrhage in ≥ 50% of the total lesion area or who have a hemorrhage in the subfoveal region of the study eye and in whom the hemorrhage area is ≥ 1 optic disk area
6. Subjects with vitreous hemorrhage in the study eye
7. Subjects who have undergone vitrectomy
8. Subjects with a history of retinal detachment, congenital disease, or treatment and/or surgical history for retinal detachment
9. Subjects with scarring, fibrosis, or atrophy involving the center of the fovea of the study eye
10. Subjects with choroidal neovascularization in the study eye due to causes other than nAMD (however, polypoidal choroidal vasculopathy (PCV) can be enrolled)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in central retinal thickness (CRT) | Week 12
  Change in central retinal thickness (CRT) measured by OCT at Week 12 compared to baseline.

SECONDARY OUTCOMES:
Change in BCVA | Weeks 4, 8, 12
  Change in BCVA at Weeks 4, 8, and 12 compared to baseline.
Change Proportion (%) in BCVA | Weeks 4, 8, 12
  Proportion (%) of subjects showing improvement in visual acuity of ≥ 1 line (5 letters on the ETDRS chart), ≥ 2 lines (10 letters on the ETDRS chart), and ≥ 3 lines (15 letters on the ETDRS chart) at Weeks 4, 8, and 12 weeks from baseline
Proportion (%) of subjects with complete disappearance of intraretinal and subretinal fluid | Weeks 4, 8, 12
  Proportion (%) of subjects with complete disappearance of intraretinal and subretinal fluid confirmed by OCT at Weeks 4, 8, and 12 weeks compared to baseline
Proportion (%) of subjects who received rescue medication | Weeks 4, 8, 12
  Proportion (%) of subjects who received rescue medication (anti-VEGF drug) at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Kyu Hyeong Park, Study Chair — Seoul National University HospitalSeoul National University Hospital; JaeHui Kim, Principal Investigator — Kim's Eye Hospital; Iksoo Byon, Principal Investigator — Pusan National University Hospital; Min Sagong, Principal Investigator — Yeungnam University Hospital; Dong Geun Kim, Principal Investigator — Inje University
Locations (5):
- South Korea (5):
  - Busan Paik Hospital, Inje University, Busan
  - Pusan National University Hospital, Busan
  - Yeungnam University Medical Center, Daegu
  - Kim's Eye Hospital, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Specify the Plan to Share IPD: All outcome data, including anonymized individual participant data, will be shared.
  What IPD Will Be Shared: Demographic information of participants, primary outcome data, secondary outcome data, analysis code, etc.
  When Will IPD Be Available: Data will be shared starting 6 months after the trial ends and will be available for at least 5 years.
  Under What Conditions Will IPD Be Shared: Data will be available for research purposes only and will be provided to approved researchers.
  How to Access the Shared IPD: Researchers must submit a data access request form. Access to the data will be granted upon approval of the request.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will be shared starting 6 months after the trial ends and will be available for at least 5 years.
Access Criteria: Data will be available for research purposes only and will be provided to approved researchers. Researchers must submit a data access request form that includes the research objectives and methodology. Access will be granted upon approval by the data sharing committee.